CLINICAL TRIAL: NCT05721664
Title: Effect of Evidence-based Nursing Practices Training Program on the Competency of Nurses Caring for Mechanically Ventilated Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sameh Elhabashy, Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: EBNPTP-NC-MVP
Record Dates: First submitted 2023-02-01; First posted 2023-02-10 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Nursing Caries; Practice Nurse's Scope; Competence
MeSH Terms: interventions — Nurses

STUDY DESIGN:
Intervention Model Description: A prospective, true experimental, and comparative research design will be used in the current study. The type of true experiment that will be conducted is (pretest-posttest control). The study will compare the current traditional in-service training with developed (EBNTP) regarding the care of mechanically ventilated patients. True-experiment is research design where the researcher initiates an experimental treatment, randomly assigns test units and treatments to the experimental group, and use of control group
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Evidence-based nursing practices training program (Experimental): Evidence-based nursing practices training program for nurses caring mechanically ventilated patients
  Interventions: Other: Trianing program for nurse in how to provide evidence based practices for mechanically Ventilated Patients
- control group taking the traditional education (Active Comparator): control group taking the traditional education related to caring of mechanically ventilated patients
  Interventions: Other: Trianing program for nurse in how to provide evidence based practices for mechanically Ventilated Patients

INTERVENTIONS:
Other: Trianing program for nurse in how to provide evidence based practices for mechanically Ventilated Patients — Short Name: (EBNPTP) for Caring of Mechanically Ventilated Patients in terms of standardized care.
  Duration: Two weeks A number of Contact Hours: 30 hrs. associated arm (interventional arm): for study group of ICU Nurses working at National Hepatology and Tropical Medicine Research Institute (NHTMRI)
  Other Names: nursing practices guidleness

SUMMARY:
the overall aim of this study is to examine the effect of adapted Evidence-based nursing practices training program on the competency level of nurses caring for Mechanically ventilated patients in selected ICU in Egypt.

Significant of the study:

The current study is expected to improve the nurses' practices regarding caring for mechanically ventilated patients in terms of optimal quality of care by keeping them up to date with the latest (EBP). Also, it is likely to enhance nurses' confidence and work satisfaction. Accordingly, all mentioned expected outputs will significantly impact either patients or the Healthcare Delivery System (HDS) in Egypt. The implementation of the study will be expected to positively impact minimizing mortality, morbidity, length of stay, incidence of readmission, and costs. Accordingly, all mentioned expected outputs will significantly impact either patients or the Healthcare Delivery System (HDS) in Egypt. Also increases the satisfaction of patients and their families. Also, the current study is expected to encourage health care providers in Egypt to increase the engagement of EBP as a concept in patient care since EBP is rarely adopted in health care facilities especially in Egypt [21-23]. in addition to recognizing the factors that may affect the implementation of EBP in such Egyptian hospitals.

Hypothesis: H1: Nurses who are given an evidence-based nursing practices training program (μ1) demonstrate a sustainable higher change in their level of competency than those who take the current traditional in-service education (μ2) in respect of caring for mechanically ventilated patients. (H1: μ1 > μ2).

Research Design:

A prospective, true experimental, and comparative research design will be used in the current study. The type of true experiment that will be conducted is (pretest-posttest control). The study will compare the current traditional in-service training with developed (EBNTP) regarding the care of mechanically ventilated patients. True-experiment is research design where the researcher initiates an experimental treatment, randomly assigns test units and treatments to the experimental group, and use of control group [27].

Sample and Setting

The research will take place in an adult intensive care unit (ICUs) of the National Hepatology and tropical medicine research institute (NHTMRI), Cairo, Egypt. In this study, the sample size is expected to be 80 critical care nurses working in selected (ICUs) estimated by (G Power analysis). Two groups will be selected randomly from the overall sample size (study and control). All nurses should have met the following requirements to be included:

* Willing to take part in this research.
* Hold the existing position for at least three months.
* Two years or more of critical care experience.
* Nurses who intend to leave their jobs four months from now will not be eligible.

DETAILED DESCRIPTION:
Background:

Evidence-based practices (EBP) is a universal key approach for delivering standardized care using the latest evidence to enhance healthcare quality and patient outcomes. EBP is a problem-solving method to make a clinical decision within healthcare setting. Nurses play a significant role in optimizing health service productivity. Further, they directly interact with patients, especially in Intensive Care Units (ICU). Hence, healthcare organizations should always work to make it simple for nurses on the frontlines to use the best evidence in their everyday practices.

EBP in healthcare is not conceptually new. From a nursing perspective, Florence Nightingale pioneered the concept of using research evidence to dictate care. The concept of EBP changed as the nursing profession evolved, as with any other applied science. As early as 1972, British medical researcher Archibald L. Cochrane criticized the medical discipline for providing management that lacked proof by evidence. Cochrane Center, which ultimately resulted in the founding of the Cochrane Collaboration in 1993. Cochrane continues to offer systematic evaluations of randomized controlled trials of medical management to assess the efficacy of provided care. The first detailed description of EBP and nursing in primary care was published in 1996 . EBP in nursing has continue tremendous growth in the past few decades.

ICU is the department that cares for critically ill patients with severe or life-threatening illnesses, requiring constant care, close supervision, and high-alert caregivers. For critically ill patients, mechanical ventilation (MV) is the most often employed therapeutic treatment modality. MV is a machine that helps a patient breathe better when they cannot breathe effectively. Mechanically ventilated patients are suspected of developing several complications that negatively affect patient outcomes, such as increased patient costs, length of stay, morbidity, and mortality rate.

While, EBP provides opportunities for nursing practices to be more individualized and effective, one of the main obstacles in the clinical context worldwide is turning the evidence into practice. Several of these obstacles were investigated such as lack of administrative support, deficiency of interest, negative beliefs, attitudes and values, heavy patient workloads, lack of resources, or inadequate staffing. By 2020, according to the Institute of Medicine (2009), 90% of clinical decisions should be supported by evidence.

Since, EBP has been acknowledged as one of the fundamental skills that clinical nurses should possess. Nurses alleged that there was a worldwide issue with having insufficient EBP knowledge and skills for using EBP in practice. Nurses in Egypt has no exception, several studies recommended extensive training of the nurses due to inadequate nurses' practices regarding caring for patients with MV . Since, healthcare is rapidly evolving and there are no shortcuts of practices, peak performance requires a lifelong passion of learning to guarantee that the patients receive the best care in term of EBP as a priority globally. Hence, the overall aim of this study is to examine the effect of adapted Evidence-based nursing practices training program on the competency level of nurses caring for Mechanically ventilated patients in selected ICU in Egypt.

Significant of the study:

The current study is expected to improve the nurses' practices regarding caring for mechanically ventilated patients in terms of optimal quality of care by keeping them up to date with the latest (EBP). Also, it is likely to enhance nurses' confidence and work satisfaction. Accordingly, all mentioned expected outputs will significantly impact either patients or the Healthcare Delivery System (HDS) in Egypt. The implementation of the study will be expected to positively impact minimizing mortality, morbidity, length of stay, incidence of readmission, and costs. Accordingly, all mentioned expected outputs will significantly impact either patients or the Healthcare Delivery System (HDS) in Egypt. Also increases the satisfaction of patients and their families. Also, the current study is expected to encourage health care providers in Egypt to increase the engagement of EBP as a concept in patient care since EBP is rarely adopted in health care facilities especially in Egypt. in addition to recognizing the factors that may affect the implementation of EBP in such Egyptian hospitals.

Hypothesis: H1: Nurses who are given an evidence-based nursing practices training program (μ1) demonstrate a sustainable higher change in their level of competency than those who take the current traditional in-service education (μ2) in respect of caring for mechanically ventilated patients. (H1: μ1 > μ2).

Conceptual Framework:

The revised Johns Hopkins Evidence-Based Practice (JHEBP) Model for Nurses (2020) is designed as a systematic and efficient approach to EBP in nursing that helps solve problems. Since a conceptual framework illustrates the underlying structure and how researchers think their study will operate, (JHEBP) model encompasses three essential components: Inquiry, Practice, and Learning

Inquiry:

Inquiry is a basis for healthcare practice and incorporates a deliberate effort to question, examine, and gather information about faced problem through clinical observation, assessment, and composed experience within the clinical setting. The stated inquiry of the current study is indicated by the researchers' observation, experience, and previous research. Moreover, a pre-assessment of the nurses' level of competency may confirm the study inquiry.

Practice Practice demonstrates how nurses apply their knowledge to their work. It consists of three items' process (Practice Question, Evidence, and Translation), it is the who, when, where, what, why, and how that demonstrates the range of clinical activities that shape the provided care. In order to JHEBP PET process, the researcher formulated the following PET process

Learning:

learning defined by Braungart et al. (2014) as "a reasonably permanent change in skill, and/or behavior as a result of experience". Transformational learning, also known as behavioral changes, the basic objective of learning is to keep nurses' behavior from changing. Staff must believe that changing practice will enhance the standard of care and have a positive impact on patients' lives for EBP to be properly embraced and integrated into the organization.

Research Design:

A prospective, true experimental, and comparative research design will be used in the current study. The type of true experiment that will be conducted is (pretest-posttest control). The study will compare the current traditional in-service training with developed (EBNTP) regarding the care of mechanically ventilated patients. True-experiment is research design where the researcher initiates an experimental treatment, randomly assigns test units and treatments to the experimental group and uses of control group.

Sample and Setting

The research will take place in an adult intensive care unit (ICUs) of the National Hepatology and tropical medicine research institute (NHTMRI), Cairo, Egypt. In this study, the sample size is expected to be 80 critical care nurses working in selected (ICUs) estimated by (G Power analysis). Two groups will be selected randomly from the overall sample size (study and control). All nurses should have met the following requirements to be included:

* Willing to take part in this research.
* Hold the existing position for at least three months.
* Two years or more of critical care experience.
* Nurses who intend to leave their jobs four months from now will not be eligible.

Study variables and measured outcomes:

Evidence-Based Nursing Training Program (EBNTP) regards caring for mechanically ventilated patients (independent variable). It's an integrated training clinical course designed by the researchers in terms of the concept of EBP. It consists of eight domains: Minimize ventilator exposure, provide oral hygiene care; management of subglottic secretion; ensure adequate staffing, Bronchial hygiene maneuvers, change ventilator circuits; give the prescribed medications recommended in the VAP bundle; and promote extubation and MV liberation. Nurses' level of competency is the dependent variable and measured outcome of the current experiment that will be assessed by a structured observational (EBNCAC).

. Tools of Data Collection: For the purpose of the study, only one adapted data collection tool will be used. "Evidence-Based Nursing Competency Assessment Checklist (EBNCAC) concerned with caring of MV patients" is a structured observational checklist that was adapted and compiled from many resources, including the Cochrane Library, AACN, and American Association for Respiratory Care (AARC). Critical nursing and medical experts reviewed the tool for content validity. Additionally, the program was adjusted to take advantage of the setting amenities.

The charge nurses in the chosen ICU will serve as the assessors, who will observe and assess the nurses' performance while caring the MV patients. Background information on the participants will also be gathered, including participant code number, sex, years of ICU experience, staff category, and educational level.

The eight domains encompassed in the training program were covered in the tool and transformed into specific nursing actions. It consists of 74 points. Nursed response to each item will be graded on a scale of 2 to 0. An item that is done correctly and satisfactorily by the nurse will receive a score of 2; handled unsatisfactory item will get 1, Items that are not performed will receive a zero score. The perceived level of skill will be classified into three categories based on the total score of 148: High (> 120 / >80%), Moderate (74-120 / 50-80%), and Low (74 / 50%).

Procedure:

The study will be carried out in three stages: planning and design, empirical, and evaluation & follow-up. The planning and design phase will involve a recent review of relevant literature, the creation of the structured study tool, the formulation of integrated training program content in light of EBP, and prepare the teaching materials related to caring for MV patients while taking into consideration the qualifications of targeted nurses and the facilities in the selected setting. The educational tool and its content will be revised by medical and nursing specialists to assure their content validity. Additionally, prior to beginning the implementation phase, official approval and ethical approval will be requested.

The empirical phase will be implemented in two stages once official permission and ethical approval are given to proceed with the proposed study:

The first stage will begin by randomly assigning the selected nurses to two paired groups (study and control) 40 nurses each. The nurses in the control group are those who are taking the current traditional in-service education (It is a daily, unstructured training sessions given in clinical settings regarding caring for ICU patients). Another group will be taking the EBNTP (study group). The second stage will begin with the selected ICU charge nurses administering the study's pre-assessment for the study and control group in real clinical settings using the study tool (EBNCAC). Following that, the recommended EBNTP will be administered to the study group for one week, while the control group receives the previously mentioned traditional in-service education.

Once empirical is complete, the 3rd phase will be initiated by evaluation & follow-up. It will include immediate 1st post-assessment for the study and control group of nurses that will measure the change expected to happen directly at the end of the program. Follow-up (2nd post-assessment) will be started one month later, followed by 3rd post-assessment after three months from the end of the EBNTP. 2nd and 3rd post-assessments aimed to measure the sustainability of the change in the level of competency of nurses. In fact, the nurses consider that they have learned if a sustainable, permanent change in their competency has been observed.

After the empirical phase is finished, the third phase will begin with evaluation & follow-up. It will include a first post-assessment that will be conducted immediately after the program ends for both the study's nurses and the control group. The second post-assessment for follow-up will begin one month later, and the third post-assessment will begin three months after the EBNTP has ended. The purpose of the second and third post-assessments was to measure the sustainability of the change in the level of competency of nurses. The nurses actually believe that they have learned if there has been a noticeable, sustainable, and permanent change in their competency.

Finally, in response to the aim of the study, the researcher will compare the scores of the study group of nurses with the scores of the control group, which will be considered as baseline data to determine the effect of given EBNTP.

Ethical Consideration:

The proposed study will only be carried out with official approval from the ethics committee. Additionally, participation in the study is entirely optional, and each subject is free to leave at any time. The subjects' informed consent will be acquired. Through the coding of all data, the confidentiality and anonymity of the subjects are ensured; subjects are given the assurance that their data won't be used in another study without their consent, that they'll only be used for the research, and that the entire required sample in the study will be followed until it's been analyzed. All information obtained will be kept private and will not in any way influence their annual evaluation.

Data analysis The statistical package for social sciences (SPSS), version 21, will be used to enter, classify, tabulate, and analyze the collected data. Descriptive statistics, such as mean, standard deviation, frequency, and percentage, will be made. The study's hypotheses were put to the test using tests of significance, such as the paired and unpaired t-test, the chi-square test, and the ANOVA test. Between quantitative variables, Pearson's correlation coefficient was used. At p 0.05, a significant level was taken into account.

ELIGIBILITY:
Inclusion Criteria:

* Willing to take part in this research.
* Hold the existing position for at least three months.
* Two years or more of critical care experience.
* Nurses who intend to leave their jobs four months from now will not be eligible.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-11-16 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
competency level of nurses regards Caring for mechanically ventilated patients. | 3 months
  Nurses' level of competency is the dependent variable and measured outcome of the current experiment that will be assessed by the Evidence-Based Nursing Competency Assessment Checklist (EBNCAC), the score value ranged from (0-148), Competency level scale: High (>120 / >80%) Moderate ( 74- 120 / 50-80%) Low (< 74 / <50%) (for caring of Mechanically ventilated patients)

CONTACTS AND LOCATIONS:
Overall Officials: Basim Essa, Study Director — National Hepatology and tropical medicine research institute
Locations (1):
- Cairo University Hospital, Cairo, Egypt

REFERENCES:
- [Derived] Elhabashy S, Moriyama M, Mahmoud EIE, Eysa B. Effect of evidence-based nursing practices training programme on the competency of nurses caring for mechanically ventilated patients: a randomised controlled trial. BMC Nurs. 2024 Apr 2;23(1):225. doi: 10.1186/s12912-024-01869-1. PMID 38566049